CLINICAL TRIAL: NCT00857246
Title: Neoadjuvant Therapy of Gastric Cancer With Irinotecan, Cisplatin and Cetuximab Followed by Surgical Resection and Adjuvant Chemoradiation
Brief Title: Pre-operation Chemo and Antibody Therapy Followed by Surgical Resection and Adjuvant Chemoradiation for Gastric Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: Bristol-Myers Squibb (Industry); Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 04-72 (H12637); BMS #CA225112 (Other: Bristol-Myers Squibb)
Record Dates: First submitted 2009-03-04; First posted 2009-03-06 (Estimated); Results first posted 2015-03-13 (Estimated); Last update posted 2015-12-07 (Estimated); Status verified 2015-11

CONDITIONS: Gastric Cancer; Stomach Cancer
Keywords: stomach cancer; biologics; antibody; chemotherapy; chemoradiation; adjuvant therapy; neoadjuvant therapy; epidermal growth factor receptor; combination therapy
MeSH Terms: conditions — Stomach Neoplasms | interventions — Cetuximab; Irinotecan; Cisplatin; Surgical Procedures, Operative; Fluorouracil; Radiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Induction/ surgery/ chemoRT (Experimental): 1. Induction treatment (3 weeks/cycle x 4 cycles): Cisplatin and Irinotecan on days 1 and 8; Cetuximab on days 1, 8, and 15.
  2. Surgery (starts 3-4 weeks after induction treatment).
  3. Chemoradiation treatment (starts 4-6 weeks after surgery):
  weeks 1-19: Cetuximab on day 1 of every week; week 1: 5-FU and Leucovorin (LV) x 5 days; weeks 2-4: recovery; weeks 5-9: radiation, 150 cGy x 5 fractions/week x 5 weeks; week 5: 5-FU+ LV on days 1-4; week 9: 5-FU+ LV on days 1-3; weeks 14 and 19: 5-FU+LV x 5days
  Interventions: Drug: Cetuximab; Drug: Irinotecan; Drug: Cisplatin; Procedure: Surgery; Drug: 5-FU; Radiation: Radiation

INTERVENTIONS:
Drug: Cetuximab
  Other Names: Erbitux
Drug: Irinotecan
  Other Names: CPT-11; Camptosar
Drug: Cisplatin
  Other Names: Platinol-AQ
Procedure: Surgery
Drug: 5-FU
  Other Names: Fluorourocil
Radiation: Radiation

SUMMARY:
This study intends to evaluate the feasibility and treatment efficacy of adding an antibody blocking the epidermal growth factor (EGF) pathway to a neoadjuvant approach with proven efficacy developed at New York University.

DETAILED DESCRIPTION:
The overall objective of this study is the development of definitive treatments for patients with locally advanced gastric cancer. To this end, this trial is evaluating the feasibility and treatment efficacy of adding an antibody blocking the EGF pathway to a neoadjuvant approach with proven efficacy developed at New York University (NYU). The combination of Irinotecan and Cisplatin has been shown to be synergistic and active against gastric carcinoma. This trial therefore builds upon NYU previous experience with the neoadjuvant administration of Irinotecan combined with Cisplatin as well as the reported enhanced activity of Irinotecan, Cisplatin and External beam radiation when combined with Cetuximab to develop a novel neoadjuvant and adjuvant approach for the treatment of gastric and gastro-esophageal junction (GEJ) cancers. The program includes: 1) systemic combination of Irinotecan, Cisplatin and Cetuximab used as an induction, 2) followed by potentially curative gastrectomy or GEJ resection, and 3) post-operative chemoradiation as reported in the Intergroup study with the addition of Cetuximab.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have signed an approved informed consent.
* must have histologically documented untreated gastric/GEJ carcinoma (clinical stage T3 N0 or T4, or any T with N1-N3 M0)
* Patients with tumor tissue available for assessment of EGF receptor status by immuno-histochemistry (IHC).
* Patients with Performance Status 0-2.
* Patients, 18 years and older, must either be not of child bearing potential or have a negative pregnancy test within 7 days of treatment. Patients are considered not of child bearing potential if they are surgically sterile (they have undergone a hysterectomy, bilateral tubal ligation, or bilateral oophorectomy) or they are postmenopausal.
* Bone marrow function: absolute neutrophil count (ANC) at least 1,500/ul; platelets at least 100,000/ul.
* Renal function: creatinine not greater than 1.5 x institutional upper limit of normal (ULN).
* The PT and PTT should be within the range of normal values
* Hepatic function: bilirubin not greater than 1.5 x ULN; aspartate aminotransferase (AST) not greater than 2.5 x ULN.

Exclusion Criteria:

* Acute hepatitis or known HIV.
* Active or uncontrolled infection.
* Significant history of uncontrolled cardiac disease; i.e., uncontrolled hypertension, unstable angina, and congestive heart failure.
* Prior therapy that affects or targets the EGF pathway.
* Prior allergic reaction to chimerized or murine monoclonal antibody therapy or documented presence of human anti-mouse antibodies (HAMA).
* Any concurrent chemotherapy not indicated in the study protocol or any other investigational agent(s).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2005-07; Primary Completion 2011-09 (Actual); Study Completion 2015-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Theresa Ryan, MD, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Cancer Center, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: From October 2005 to November 2010, 30 patients were enrolled to the study from New York University Langone Medical Center and its affiliated hospitals.
Period: Induction Regimen
Arm/Group | Induction/ Surgery/ chemoRT
Started | 30
Completed | 27
Not Completed | 3
Not completed — Adverse Event | 1
Not completed — disease-related complications | 1
Not completed — Withdrawal by Subject | 1
Period: Surgery (Curative)
Arm/Group | Induction/ Surgery/ chemoRT
Started | 27
Completed | 21
Not Completed | 6
Not completed — disease progression | 6
Period: ChemoRT
Arm/Group | Induction/ Surgery/ chemoRT
Started | 15 (6 did not start adjuvant therapy due to disease-related complications or patient withdrawal.)
Completed | 12
Not Completed | 3
Not completed — Withdrawal by Subject | 1
Not completed — Adverse Event | 2

BASELINE CHARACTERISTICS:
Groups:
- Induction/ Surgery/ chemoRT: 1. Induction treatment (3 weeks/cycle x 4 cycles): Cisplatin and Irinotecan on days 1 and 8; Cetuximab on days 1, 8, and 15.
  2. Surgery (3-4 weeks after induction treatment).
  3. Chemoradiation treatment (4-6 weeks after surgery):
  weeks 1-19: Cetuximab on day 1 of every week; week 1: 5-FU and Leucovorin (LV) x 5 days; weeks 2-4: recovery; weeks 5-9: radiation, 150 cGy x 5 fractions/week x 5 weeks; week 5: 5-FU+ LV on days 1-4; week 9: 5-FU+ LV on days 1-3; weeks 14 and 19: 5-FU+LV x 5days
Arm/Group | Induction/ Surgery/ chemoRT
Number analyzed (Participants) | 30
Age, Customized [Number; unit: participants]
  25-34 years | 1
  35-44 years | 1
  45-53 years | 8
  54-63 years | 12
  64-73 years | 3
  74-83 years | 5
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 23
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 13
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 11
  More than one race | 0
  Unknown or Not Reported | 2
Region of Enrollment [Number; unit: participants]
  United States | 30

OUTCOME MEASURES:

1. Primary Outcome: Clinical Response Rate of an Induction Regimen Consisting of Irinotecan, Cisplatin and Cetuximab
Description: Clinical response rate is defined as the percentage of patients who responded to the induction regimen. The response is determined based on endoscopic ultrasonography (EUS) staging pre-treatment and post-treatment, CT scans pre- and post- operatively, and initial clinical stage (based on these tests) compared with the pathologic stage. Any "down-staging" of T or N stage is considered to be a result of induction therapy and counted as a clinical response.
Time Frame: 4 months from the beginning of the induction regimen
Population: Evaluable patients (known pre-treatment clinical and post-treatment pathologic stages)
Measure: Number; unit: percentage of paticipants
Arm/Group | Induction/ Surgery/ chemoRT
Number analyzed (Participants) | 25
percentage of paticipants | 40

2. Secondary Outcome: Rate of Clearance of Nodal Involvement Among Patients Who Have Received the Induction Therapy
Description: This is defined as the percentage of patients whose nodal involvement of cancer has been cleared based on surgery results.
Time Frame: 4 months from the beginning of the induction treatment
Population: Evaluable patients (known pre-treatment clinical and post-treatment pathologic stages)
Measure: Number; unit: percentage of participants
Groups:
- Induction/ Surgery/ chemoRT: 1. Induction treatment (3 weeks/cycle x 4 cycles): Cisplatin and Irinotecan on days 1 and 8; Cetuximab on days 1, 8, and 15.
  2. Surgery (starts 3-4 weeks after induction treatment).
  3. Chemoradiation treatment ( starts 4-6 weeks after surgery):
  weeks 1-19: Cetuximab on day 1 of every week; week 1: 5-FU and Leucovorin (LV) x 5 days; weeks 2-4: recovery; weeks 5-9: radiation, 150 cGy x 5 fractions/week x 5 weeks; week 5: 5-FU+ LV on days 1-4; week 9: 5-FU+ LV on days 1-3; weeks 14 and 19: 5-FU+LV x 5days
Arm/Group | Induction/ Surgery/ chemoRT
Number analyzed (Participants) | 25
percentage of participants | 0

3. Secondary Outcome: Rate of Potentially Curative Surgery
Description: This is defined as the percentage of patients who underwent curative surgery (surgery to remove all cancerous tissue).
Time Frame: 4 months from the beginning of the induction treatment
Population: patients who underwent surgery
Measure: Number; unit: percentage of participants
Arm/Group | Induction/ Surgery/ chemoRT
Number analyzed (Participants) | 27
percentage of participants | 78

4. Secondary Outcome: Rate of "Down-staging" From Pre-operative Clinical Staging
Description: This is defined as the percentage of patients who had a reduction from T3/T4 disease.
Time Frame: 4 months from the beginning of the induction treatment
Population: Evaluable patients (known pre-treatment clinical and post-treatment pathologic stages)
Measure: Number; unit: percentage of participants
Arm/Group | Induction/ Surgery/ chemoRT
Number analyzed (Participants) | 25
percentage of participants | 53

5. Secondary Outcome: Safety of the Induction Regimen
Description: This describes the number of patients who experienced grade 3 and higher adverse events related to the regimen.
Time Frame: 4 months from the beginning of the induction
Population: Patients who had at least a dose of treatment
Measure: Number; unit: participants
Groups:
- Induction Treatment: Induction treatment (3 weeks/cycle x 4 cycles): Cisplatin and Irinotecan on days 1 and 8; Cetuximab on days 1, 8, and 15.
Arm/Group | Induction Treatment
Number analyzed (Participants) | 30
participants
  Neutrophils/granulocytes | 13
  Diarrhea | 4
  Fatigue | 3
  Rash | 3
  Leukocytes | 2
  Hypomagnesmia | 2
  Hypotension | 2
  Lymphopenia | 1
  Vomiting | 1
  Dehydration | 1
  Hypophosphatemia | 1
  Hypokelemia | 1
  Stomatitis/Pharyngitis | 1
  Febrile neutropenia | 1
  Hemoglobin | 1
  Carpopedal syndrome | 1

6. Secondary Outcome: Median Overall Survival (Induction Treatment and Curative Surgery)
Description: This is the length of time from the start of treatment that half of the patients are still alive.
Time Frame: up to 5 years
Population: Patients who completed induction treatment and underwent curative surgery
Measure: Median (Full Range); unit: months
Arm/Group | Induction/ Surgery/ chemoRT
Number analyzed (Participants) | 21
months | 35.3 [1 to 81]

7. Secondary Outcome: Median Overall Survival (Adjuvant Therpary)
Description: This is the length of time from the start of treatment that half of the patients are still alive.
Time Frame: up to 5 years
Population: Patients who received at least one cycle of adjuvant therapy
Measure: Median (Full Range); unit: months
Arm/Group | Induction/ Surgery/ chemoRT
Number analyzed (Participants) | 15
months | 39.5 [8 to 81]

ADVERSE EVENTS:
Time Frame: Up to 1 year
Description: All the adverse events (AEs) from the induction to adjuvant therapies are reported here regardless of attributions.
Arm/Group | Induction/ Surgery/ chemoRT
Serious Adverse Events (participants affected / at risk) | 15/30
Other Adverse Events (participants affected / at risk) | 30/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Induction/ Surgery/ chemoRT (N=30)
Ascites (non-malignant) (Gastrointestinal disorders) | 1
Chest pain (non-cardiac and non-pleuritic) (Cardiac disorders) | 1
Dehydration (Gastrointestinal disorders) | 2
Diarrhea patients without colostomy (Gastrointestinal disorders) | 2
Dysphagia, esophagitis, odynophagia (painful swallowing) (Gastrointestinal disorders) | 1
Fatigue (lethargy, malaise, asthenia) (General disorders) | 1
Fever (in the absence of neutropenia) (General disorders) | 2
Abdominal pain or cramping (Gastrointestinal disorders) | 1
Gastrointestinal-Other: small bowel obstruction (General disorders) | 2
Hematemesis (Gastrointestinal disorders) | 1
Hemoglobin (Blood and lymphatic system disorders) | 2
Hypotension (Cardiac disorders) | 2
Infection without neutropenia (Infections and infestations) | 2
Musculoskeletal-Other: muscle twitching (Musculoskeletal and connective tissue disorders) | 1
Neutrophils/granulocytes (ANC/AGC) (Blood and lymphatic system disorders) | 1
Syndromes-Other: carpopedal (Musculoskeletal and connective tissue disorders) | 1
Thrombosis/embolism (Vascular disorders) | 3
Vomiting (Gastrointestinal disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Induction/ Surgery/ chemoRT (N=30)
Abdominal pain or cramping (Gastrointestinal disorders) | 14
Alkaline phosphatase (Investigations) | 9
Allergic rhinitis (including sneezing, nasal stuffiness, postnasal drip) (Immune system disorders) | 1
Alopecia (Skin and subcutaneous tissue disorders) | 3
Anorexia (Gastrointestinal disorders) | 19
Arthtitis (Musculoskeletal and connective tissue disorders) | 1
Bicarbonate (Metabolism and nutrition disorders) | 3
Bilirubin (Hepatobiliary disorders) | 2
Cardiovascular/Arrhythmia-Other: Atrial Fibrillation (Cardiac disorders) | 1
Chest pain (non-cardiac and nonpleuritic (Cardiac disorders) | 2
Constipation (Gastrointestinal disorders) | 12
Cough (Respiratory, thoracic and mediastinal disorders) | 4
Creatitine (Investigations) | 1
Dehydration (Gastrointestinal disorders) | 3
Dermatology/Skin-Other: blister (Skin and subcutaneous tissue disorders) | 1
Dermatology/Skin-Other: fissurs (Skin and subcutaneous tissue disorders) | 5
Dermatology/Skin-Other: Itchy scalp (Skin and subcutaneous tissue disorders) | 1
Dermatology/Skin-Other: Paronychia (Skin and subcutaneous tissue disorders) | 2
Dermatology/Skin-Other: surgical scar stiffness (Skin and subcutaneous tissue disorders) | 1
Diarrhea patients without colostomy (Gastrointestinal disorders) | 20
Dizziness/lightheadedness (Nervous system disorders) | 7
Dry eye (Eye disorders) | 1
Dry skin (Skin and subcutaneous tissue disorders) | 7
Dyspepsia/heartburn (Gastrointestinal disorders) | 4
Dysphagia, esophagitis, odynophagia (painful swallowing) (Gastrointestinal disorders) | 6
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 5
Edema (General disorders) | 2
Fatigue (lethargy, malaise, asthenia) (General disorders) | 20
Febrile neutropenia (Blood and lymphatic system disorders) | 2
Fever (in the absence of neutropenia) (General disorders) | 4
Flatulence (Gastrointestinal disorders) | 1
Flushing (Vascular disorders) | 2
Gastritis (Gastrointestinal disorders) | 1
Gastrointestinal-Other: Abdominal bloating (Gastrointestinal disorders) | 2
Gastrointestinal-Other: Early Satiety (Gastrointestinal disorders) | 1
Gastrointestinal-Other: Hemorrhoids (Gastrointestinal disorders) | 1
Gastrointestinal-Other: Oral Lesions (Gastrointestinal disorders) | 3
Gastrointestinal-Other: Pressure discomfort (Gastrointestinal disorders) | 1
Hand-foot skin reaction (Skin and subcutaneous tissue disorders) | 3
Headache (Nervous system disorders) | 3
Hemoglobin (Blood and lymphatic system disorders) | 14
Hemorrhage/bleeding without grade 3 or 4 thrombocytopenia (Gastrointestinal disorders) | 2
Hiccoughs (hiccups, singultus) (Respiratory, thoracic and mediastinal disorders) | 1
Hyperglycemia (Metabolism and nutrition disorders) | 11
Hyperkalemia (Metabolism and nutrition disorders) | 3
Hypermagnesemia (Metabolism and nutrition disorders) | 5
Hypernatremia (Metabolism and nutrition disorders) | 1
Hypertension (Cardiac disorders) | 1
Hypoalbuminemia (Hepatobiliary disorders) | 7
Hypocalcemia (Metabolism and nutrition disorders) | 8
Hypoglycemia (Metabolism and nutrition disorders) | 4
Hypokalemia (Metabolism and nutrition disorders) | 10
Hypomagnesmia (Metabolism and nutrition disorders) | 7
Hyponatremia (Metabolism and nutrition disorders) | 6
Hypophosphatemia (Metabolism and nutrition disorders) | 5
Hypotension (Cardiac disorders) | 3
Infection without neutropenia (Infections and infestations) | 4
Insomnia (Nervous system disorders) | 3
Leukocytes (total WBC) (Blood and lymphatic system disorders) | 14
Lymphopenia (Blood and lymphatic system disorders) | 10
Mood alteration-depression (Nervous system disorders) | 1
Mouth dryness (Gastrointestinal disorders) | 1
Nail changes (Skin and subcutaneous tissue disorders) | 2
Nausea (Gastrointestinal disorders) | 24
Neuropathy-sensory (Nervous system disorders) | 3
Neutrophils/granulocytes (ANC/AGC) (Blood and lymphatic system disorders) | 21
Ocular/Visual - Other: periorbital edema (Eye disorders) | 1
Pain-Other: back pain (Musculoskeletal and connective tissue disorders) | 2
Pain-Other: cramps (Musculoskeletal and connective tissue disorders) | 1
Pain-Other: heels (Musculoskeletal and connective tissue disorders) | 1
Pain-other: incision site (Injury, poisoning and procedural complications) | 5
Pain-other: thigh pain (Musculoskeletal and connective tissue disorders) | 1
Pain-Other: toungue (Gastrointestinal disorders) | 1
Palpitations (Cardiac disorders) | 1
Platelets (Blood and lymphatic system disorders) | 13
Pleural effusion (non-malignant) (Respiratory, thoracic and mediastinal disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1
Pulmonary-Other: sputum (Respiratory, thoracic and mediastinal disorders) | 1
Radiation dermatitis (Skin and subcutaneous tissue disorders) | 1
Rash/dermatitis associated with high-dose chemotherapy or BMT studies. (Skin and subcutaneous tissue disorders) | 7
Rash/desquamation (Skin and subcutaneous tissue disorders) | 24
Rigors, chills (General disorders) | 4
SGOT (AST) (serum glutamic oxaloacetic transaminase) (Hepatobiliary disorders) | 6
SGPT (ALT) (serum glutamic pyruvic transaminase) (Hepatobiliary disorders) | 7
Sinus Tachycardia (Cardiac disorders) | 1
Stomatitis/pharyngitis (oral/pharyngeal mucositis) (Gastrointestinal disorders) | 6
Sweating (diaphoresis) (General disorders) | 2
Taste disturbance (dysgeusia) (Gastrointestinal disorders) | 4
Thrombosis/embolism (Vascular disorders) | 1
Vision-blurred vision (Eye disorders) | 1
Voice changes/stridor/larynx (e.g., hoarseness, loss of voice, laryngitis) (Respiratory, thoracic and mediastinal disorders) | 2
Vomiting (Gastrointestinal disorders) | 12
Weight gain (General disorders) | 1
Weight loss (General disorders) | 16
Wound-infectious (Skin and subcutaneous tissue disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes